CLINICAL TRIAL: NCT00328913
Title: Effectiveness of 5-Hydroxytryptophan on Satiety in a Randomised, Placebo Controlled, Time Blinded Study, in Overweight Women
Brief Title: The Effect of 5-Hydroxytryptophan (5-HTP) on Satiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Laboratoire Oenobiol (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P6880
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Obesity
Keywords: satiety; food intake; mood; wellness; weight management
MeSH Terms: conditions — Obesity | interventions — 5-Hydroxytryptophan; Dietary Supplements

INTERVENTIONS:
Drug: 5-hydroxytryptophan (food supplement)

SUMMARY:
The aim of the study is to show evidence of the efficacy of 5-HTP to induce satiety and to reduce food intake (confirmatory study).

The primary objective of the present study is to determine:

* the effectiveness of a 5-HTP preparation on satiety markers (before intake of a meal and during the day)

The secondary objectives of the present study are to determine the effectiveness of a 5-HTP preparation on:

* food consumption (amount and composition) during a free meal (dinner);
* wellness after one week supplementation;
* the intermeal interval;
* body weight and waist-hip ratio (WHR).

DETAILED DESCRIPTION:
One of the physiological factors regulating the food intake pattern is satiety. Satiety is defined as the absence of ingestive motivation, which ends when the next meal is initiated (Blundell et al., 1996). Food intake affects a number of physiological objective parameters in blood known to be involved in signalling satiety, such as glucose (Melanson et al, 1999; Chapman et al, 1999; Campfield et al, 1996), insulin (Speechly et al, 2000) and cholecystokinin (CCK) (Gutzwiller et al., 2000; Beglinger et al., 2001; French et al., 2000; Degen et al., 2001; Burton-Freeman et al., 2002, 2004). More recently, the gastric hormone ghrelin was identified as a marker for hunger and meal initiation (De Graaf et al., 2004).

Humans do not only eat in response to a metabolic or physiological need. Humans also respond to a significant extent to other internal subjective and emotional signals (clues). The exact relations between the physiological internal signals and subjective and emotional internal signals are not known. Besides also external and social factors modulate physiological-derived hunger and satiety signals.

Though the regulation of food intake has been studied quite extensively, the underlying mechanism is not elucidated yet and still new factors involved in this regulation are being found. It is known that the macronutrients such as lipids, proteins and carbohydrates affect satiety differently, but this mechanism is still not very clear either.

Nowadays, more and more food supplements become available suggesting to affect hunger and satiety sensations, resulting in the long-term in weight loss. For example dietary fibres are known for their satiating effect.

The food supplement 5-HTP is used for this purpose as well. The food supplement, already available in the United States and in Italy, has been investigated for multiple indications such as migraine, depression, anxiety, fibromyalgia, hypertension, insomnia and obesity.

Different clinical studies have been performed with 5-HTP for more than three decades now. With respect to lowering of food intake, 5-HTP has been studied as well.

5-HTP is an amino acid produced by the human body from the essential amino acid L-tryptophan, which is found in food products. Its clinical value is the ability to increase production of serotonin. As a potentially valuable supplement it has been used clinically for more than 30 years. 5-HTP occurs naturally in two places - the human body and the seeds of the Griffonia simplicifolia, a West African medicinal plant.

5-HTP is the amino acid precursor of serotonin. Normal levels of serotonin are important for emotional well-being, may play a role in appetite suppression, and decreased carbohydrate and fat intake. Only free plasma tryptophan can cross the blood brain barrier via a carrier protein to enter the central nervous system (CNS). Once in the CNS, tryptophan is converted to 5-HTP and then is decarboxylated to serotonin. The levels, and possible function, of several neurotransmitters can be influenced by the supply of their dietary products. A reduction in tryptophan has been correlated to a reduction in serotonin (Curcio et al., 2005).

The 5-HTP metabolism is then influenced by plasma tryptophan levels, which are related to food intake. Serotonin synthesis is directly dependent on the availability of the specific precursor tryptophan and on the nutritional status.

The effect of 5-HTP intake on food intake and mood is based on the serotonin production. Numerous studies have shown that long-term consumption of 5-HTP (levels up to 900 mg daily) reduced food intake and resulted in weight loss.

In a previous study by Laboratoire Oenobiol with moderately overweight men aged 20-40 years, given 50 or 150 mg 5-HTP half an hour before lunch and half an hour before dinner, a reduced energy intake with 300 mg 5-HTP compared to placebo was found. This was supplied acutely on one day.

The study reported a linear dose related effect, with significant food intake inhibition effect with a 300 mg/day 5-HTP dose. The dose of 100 mg/day did not produce statistically significant effects compared to placebo. However, 100 mg of 5-HTP could prove to be sufficient if given under chronic administration conditions.

In the present study therefore subjects will be supplied with 100 mg 5-HTP daily for one week. Hunger and satiety feelings, food intake and wellness will be investigated. The study will be conducted with overweight women, assuming that this group of subjects will be the target group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by:

   * The TNO health and lifestyle questionnaire
   * Physical examination
2. Females aged 18 through 65 years on Day 01 of the study
3. Body mass index (BMI) 25 - 32 kg/m2 (if enough subjects are available, subjects with a BMI 25 - 30 kg/m2 will be included first).
4. Regular and normal Dutch eating habits (consuming mostly three main meals including breakfast) as assessed by the questionnaire on health and lifestyle
5. Non-restraint eaters, defined by a score of < 3.4 on the Dutch Eating Behaviour Questionnaire
6. Using oral contraceptives for > 3 months (only fixed phase)
7. Voluntary participation
8. Having given written informed consent
9. Willing to comply with the study procedures
10. Willing to agree to the use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
11. Willing to agree to the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from participation:

1. Participation in any clinical trial including blood sampling and/or administration of pharmaceutical or nutritional substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including blood sampling and/or oral, intravenous, or inhalatory administration of pharmaceutical or nutritional substances
3. Mental status that is incompatible with the proper conduct of the study (including depression)
4. Having a history of medical or surgical events that may significantly affect the study outcome, including metabolic or endocrine disease, especially diabetes type I or II; cardiovascular diseases (including hypertension); gastrointestinal diseases, including events that affect nutrient uptake or appetite; or using medication that may interfere with 5-HTP (antidepressants [selective serotonin reuptake inhibitors {SSRIs}, monoamine oxidase inhibitors {MAOIs}], migraine medication, or some hypertension medication).
5. Smoking
6. Having a history of drug abuse
7. Claustrophobia
8. Alcohol consumption > 21 units (glasses)/week
9. Not willing to stop use of supplements of minerals or vitamins from screening onwards
10. Reported food allergy or sensitivity (wheat, milk, eggs, nuts, etc.)
11. Reported unexplained weight loss or weight gain of > 2 kg in the month prior to pre-study screening
12. Practicing sports > 10 hours a week
13. Reported slimming or medically prescribed diet
14. Reported vegan, vegetarian, or macrobiotic lifestyle
15. Pregnant or lactating or wishing to become pregnant in the period of the study
16. Recent blood or plasma donation (< 1 month prior to Day 01 of the study)
17. Not willing to give up blood/plasma donation during the study
18. Personnel of TNO Quality of Life (located in Zeist), their partners and their first and second degree relatives
19. Not having a general practitioner
20. Not willing to accept information-transfer concerning participation in the study; or information regarding health, like laboratory results, findings at anamnesis or physical examination, and eventual adverse events to and from general practitioner.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-03; Study Completion 2006-07

PRIMARY OUTCOMES:
satiety scores (visual analog scores)

SECONDARY OUTCOMES:
food intake
wellness
intermeal interval
body weight and waist-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands